CLINICAL TRIAL: NCT06000683
Title: Empowering Patients' Lung Cancer Screening Uptake (Empower LCS)
Brief Title: Empowering Patients' Lung Cancer Screening Uptake
Acronym: Empower-LCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Gelareh Sadigh, Associate Professor, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 3432; UCI 23-107 (Other: University of California Irvine IRB)
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Results first posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: Patient participants (n=70) will receive the study intervention, complete surveys and a subset of them (n=11) will participate in a one-time qualitative interview.
  Provider participants (n=9) will not receive any intervention. Provider participants will participate in a one-time survey, and a subset of them (n=5) will participate in a one-time qualitative interview.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Empower LCS (Experimental): Patient will be given education material(addressing knowledge barriers); patients' referral to financial navigation resources (addressing health-related social risks); and patients' reminder to discuss LCS during PCP visit. Providers will also be notified of eligibility of their patients to receive LCS.
  Interventions: Behavioral: Patient education; Behavioral: Referral to financial navigation resources; Behavioral: Patient Reminders; Behavioral: Provider Reminers

INTERVENTIONS:
Behavioral: Patient education — Patients will be sent information (in preferred language) on lung cancer risk, lung cancer screening (LCS) benefits, harms, false positive rates, recommendations of follow-up for positive results, and exam insurance coverage.
Behavioral: Referral to financial navigation resources — Patients who self-report needing help with health-related social risks at baseline will be sent a brochure (in preferred language) from patient advocate foundation (PAF), a national non-profit financial navigation organization, where patients can self-refer.
Behavioral: Patient Reminders — Within 2 weeks prior to primary care appointment, patients will receive a text message or a phone call (if not having a phone that receives text messaging) encouraging patients to discuss the LCS with their provider.
Behavioral: Provider Reminers — Within 2 weeks prior to primary care appointment, providers will be notified of their patient's eligibility for LCS.

SUMMARY:
Lung cancer is the leading cause of cancer related mortality. Lung cancer screening (LCS) with low dose computed tomography (LDCT) decreases mortality rate of lung cancer by 20%. Yet many patients who are eligible for lung cancer screening are still falling through the cracks which prevents patients the ability to detect lung cancer early. This study will test the effect of a a multi-level intervention on ordering LDCT within 6 months after patient enrollment. Our proposed intervention includes (1) Primary care provider notifications of patients' LCS eligibility; (2) patients' education ; (3) patients' referral to financial navigation resources; and (4) patients' reminder to discuss LCS during PCP visit.

ELIGIBILITY:
Patients' Inclusion Criteria:

1. Aged 50- 80 years of age.
2. Be able to Speak English, Spanish, or Vietnamese
3. Must have a scheduled appointment with their Primary Care Providers within next one to three months.
4. The Scheduled PCP appointment is at any of the UCI Health primary care clinics in Orange County including two UCI federally qualified health centers
5. History of 20 pack year smoking history ( based on survey self report)
6. Current smoker or a former smoker who has quit smoking within the last 15 years (based on survey self report)

Patients' Exclusion Criteria:

1. Prior history of lung cancer
2. chest CT for any reason in the last 12 months based on self-report and UCI EMR
3. history of Alzheimer's disease or dementia

Providers' Inclusion Criteria:

1. Primary Care Providers whose patients were enrolled in the Empower LCS trial.
2. Received notifications about the eligibility of their patients for lung cancer screening.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2023-10-13 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gelareh Sadigh, MD, Principal Investigator — University of California, Irvine
Locations (7):
- United States (7):
  - UCI Health - Costa Mesa, Costa Mesa, California
  - UCI Health Gottschalk Medical Plaza, Irvine, California
  - UCI Health - Laguna Hills, Laguna Hills, California
  - UCI Health - Newport Beach MacArthur, Newport Beach, California
  - UCI Medical Center, Orange, California
  - UCI Health - Tustin, Tustin, California
  - UCI Health-Yorba Linda, Yorba Linda, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited via email, phone, mail or in-person outreach. 70 eligible patients consented to study and were enrolled.
  Primary care providers taking care of patient participants were recruited via email outreach. A total of 9 provider consented to the study.
Pre-assignment Details: Protocol enrollment reflects the 70 patient participants of the study who consented to study and received study intervention.
  We further reached out to primary care providers of patient participants, and 9 providers consented to study and completed a survey.
Groups:
- Patient Participants: All patients received the Empower LCS intervention, including: (1) a decision aid; (2) text reminder to encourage LCS discussion with primary care providers (PCPs); (3) PCP notifications on eligibility and barriers, and (4) financial hardship and health-related social needs support.
- Provider Participants: Primary care providers taking care of Empower LCS patient participants
Period: Overall Study
Arm/Group | Patient Participants | Provider Participants
Started | 70 | 9
Completed | 70 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patient Participants | Provider Participants | Total
Number analyzed (Participants) | 70 | 9 | 79
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 70 | 9 | 79
Perceived risk of lung cancer [Mean (Standard Deviation); unit: scores on a scale] — 3-item question with responses using 5-point Likert scale (score range: 3-15); higher score = higher perceived risk of lung cancer Population: This variable is only measured for patient participants.
  scores on a scale
    number analyzed (Participants) | 70 | 0 | 70
    (all) | 9.9 (3) |  | 9.9 (3)
Perceived severity of lung cancer [Mean (Standard Deviation); unit: scores on a scale] — 5-item question with responses using 5-point Likert scale (score range: 5-25); higher score = higher perceived severity of lung cancer Population: This variable is only measured for patient participants.
  scores on a scale
    number analyzed (Participants) | 70 | 0 | 70
    (all) | 16.3 (2.7) |  | 16.3 (2.7)
Perceived benefits of LCS [Mean (Standard Deviation); unit: scores on a scale] — 6-item question with responses using 5-point Likert scale (score range: 6-30); higher score = higher perceived benefits of LCS Population: This variable is only measured for patient participants.
  scores on a scale
    number analyzed (Participants) | 70 | 0 | 70
    (all) | 24.6 (3.5) |  | 24.6 (3.5)
Perceived barriers of LCS [Median (Standard Deviation); unit: scores on a scale] — 19-item question with responses using 5-point Likert scale (score range: 19-95); higher score = higher perceived barriers of LCS Population: This variable is only measured for patient participants.
  scores on a scale
    number analyzed (Participants) | 70 | 0 | 70
    (all) | 40.7 (14.4) |  | 40.7 (14.4)
Self- efficacy for LCS [Mean (Standard Deviation); unit: scores on a scale] — 10-item question with responses using 5-point Likert scale (score range: 10-50); higher score = higher perceived self-efficacy for LCS Population: This variable is only measured for patient participants.
  scores on a scale
    number analyzed (Participants) | 70 | 0 | 70
    (all) | 40.4 (6.3) |  | 40.4 (6.3)
Perceived Knowledge of LCS [Mean (Standard Deviation); unit: scores on a scale] — 8-item question scored by awarding one point per correct answer selected and one point per incorrect answer not selected. The score was calculated as sum of all points (score range 0-8); higher score = higher knowledge of LCS Population: This variable is only measured for patient participants.
  scores on a scale
    number analyzed (Participants) | 70 | 0 | 70
    (all) | 1.9 (1) |  | 1.9 (1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Male | 50 | 0 | 50
  Sex: Female | 20 | 0 | 20
  Sex: Unknown/not collected | 0 | 9 | 9
Age, Customized [Count of Participants; unit: Participants]
  Age: <50 yrs old | 0 | 6 | 6
  Age: 50-59 yrs old | 21 | 2 | 23
  Age: 60-69 yrs old | 40 | 1 | 41
  Age: +70 yrs old | 9 | 0 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 13 | 5 | 18
  Race: Black | 1 | 0 | 1
  Race: Other | 25 | 2 | 27
  Race: White | 31 | 2 | 33

OUTCOME MEASURES:

1. Primary Outcome: Order of LDCT
Description: Number of participants who were ordered screening with Low Dose Computed Tomographyorder (LDCT) within 6 months after enrollment, assessed with self-reported surveys or EMR data extraction.
Time Frame: within 6 months of enrollment
Population: The outcome is being reported among all 70 enrolled patient participants based on data available through 6-months follow-up survey or EMR.
Measure: Count of Participants; unit: Participants
Arm/Group | Patient Participants
Number analyzed (Participants) | 70
Participants | 50

2. Secondary Outcome: Receipt of LDCT
Description: Number of participants who were completed screening with Low Dose Computed Tomographyorder (LDCT) within 6 months after enrollment, assessed with self-reported surveys or EMR data extraction.
Time Frame: Within 6 months of enrollment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Empower LCS
Number analyzed (Participants) | 70
Participants | 17

3. Secondary Outcome: LCS Discussion
Description: Number of participants who had a discussion about screening with Low Dose Computed Tomographyorder (LDCT) with their primary care provider measured within 6 months after enrollment, through self-reported surveys or EMR documentation of discussion in the primary care notes.
Time Frame: within 6 months after enrollment
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Empower LCS
Number analyzed (Participants) | 70
Participants | 43

4. Secondary Outcome: Perceived Risk of Lung Cancer
Description: 3-item validated survey questions (from Carter Harris et al) assessing patients' perceived risk of lung cancer. Item responses use 5-point Likert scale. Total scores are calculated by summing item responses. Score is ranging between 3-15. Higher score= higher perceived risk of lung cancer.
Time Frame: At 6 months post-enrollment
Population: This outcome is measured only among participants who completed the 6-months follow-up survey.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Empower LCS
Number analyzed (Participants) | 42
scores on a scale | 10.1 (3)

5. Secondary Outcome: Perceived Severity of Lung Cancer
Description: 5-item validated survey questions assessing patients' perceived severity of lung cancer. Item responses use 5-point Likert scale. Total scores are calculated by summing item responses. Score is ranging between 5-25. Higher score= higher perceived severity of lung cancer.
Time Frame: At 6 months post-enrollment
Population: This outcome is measured only among participants who completed the 6-months follow-up survey.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Empower LCS
Number analyzed (Participants) | 42
scores on a scale | 18.1 (3.1)

6. Secondary Outcome: Perceived Benefit of Lung Cancer Screening
Description: 6-item validated survey questions (from Carter Harris et al) assessing patients' perceived benefits of lung cancer screening. Item responses use 5-point Likert scale. Total scores are calculated by summing item responses. Score is ranging between 6-30. Higher score= higher perceived benefits of lung cancer screening.
Time Frame: At 6 months post-enrollment
Population: This outcome is measured only among participants who completed the 6-months follow-up survey.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Empower LCS
Number analyzed (Participants) | 42
scores on a scale | 24.7 (4.7)

7. Secondary Outcome: Perceived Barriers to Lung Cancer Screening
Description: 19-item validated survey questions (from Carter Harris et al) assessing patients' perceived barriers to lung cancer screening. Item responses use 5-point Likert scale. Total scores are calculated by summing item responses. Score is ranging between 19-95. Higher score= higher perceived barriers to lung cancer screening.
Time Frame: At 6 months post-enrollment
Population: This outcome is measured only among participants who completed the 6-months follow-up survey.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Empower LCS
Number analyzed (Participants) | 42
scores on a scale | 37.5 (15.6)

8. Secondary Outcome: Perceived Self-efficacy for Lung Cancer Screening
Description: 10-item validated survey questions (from Carter Harris et al) assessing patients' perceived self-efficacy to undergo lung cancer screening. Item responses use 5-point Likert scale. Total scores are calculated by summing item responses. Score is ranging between 5-50. Higher score= higher perceived self-efficacy.
Time Frame: At 6 months post-enrollment
Population: This outcome is measured only among participants who completed the 6-months follow-up survey.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Empower LCS
Number analyzed (Participants) | 42
scores on a scale | 41.7 (7.5)

9. Secondary Outcome: Knowledge About Lung Cancer and Screening
Description: Knowledge of lung cancer and LCS was assessed using 8-items validated questions (from Volk et al), and scored by awarding one point per correct answer selected and one point per incorrect answer not selected. The total score was calculated as sum of all points. Total score ranged between 0 to 8. Higher score= higher knowledge.
Time Frame: At 6 months post-enrollment
Population: This outcome is measured only among participants who completed the 6-months follow-up survey.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Empower LCS
Number analyzed (Participants) | 42
scores on a scale | 2.7 (1.6)

10. Secondary Outcome: Providers' Perceived Barriers to Lung Cancer Screening
Description: 9-item survey questions assessing providers' perceived barriers to lung cancer screening. Item responses use 5-point Likert scale. Total scores are calculated by summing item responses. Score is ranging between 9-45. Higher score= higher perceived barriers to lung cancer screening.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Primary Care Providers: Providers taking care of Empower LCS patient participants
Arm/Group | Primary Care Providers
Number analyzed (Participants) | 9
Score on a scale | 24.1 (4.2)

11. Other Pre Specified Outcome: Patient and Provider Experience With Intervention
Description: Patient and Providers were asked questions about their experience with intervention components. Outcomes
Time Frame: At the end of all study enrollments a subgroup of patients and providers were interviewed
Population: A subsample of patients and providers were recruited to participate in qualitative interviews. Each row summarizes a theme identified in thematic analysis. The number of participants that endorsed/discussed the theme are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Empower LCS | Primary Care Providers
Number analyzed (Participants) | 11 | 5
Participants
  Shared Positive Views of Current Lung Cancer Screening Protocols | 4 | 2
  Shared Negative Views of Current Lung Cancer Screening Protocols | 3 | 4
  Identified Barriers to Lung Cancer Screening | 6 | 5
  Shared Impact of Intervention | 8 | 5
  Provided Suggestions for Future Trials | 8 | 4

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 6 months
Arm/Group | Patient Participants | Provider Participants
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/9
Other Adverse Events (participants affected / at risk) | 0/70 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-02): https://cdn.clinicaltrials.gov/large-docs/83/NCT06000683/Prot_SAP_000.pdf